CLINICAL TRIAL: NCT03548779
Title: North Carolina Genomic Evaluation by Next-generation Exome Sequencing, 2
Acronym: NCGENES2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); East Carolina University (Other); Mission Health System, Asheville, NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17-0816; U01HG006487 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy; Seizure; Neuromuscular Diseases; Brain Malformation; Intellectual Disability; Autism Spectrum Disorder; Hypotonia; Inborn Errors of Metabolism; Movement Disorders; Genetic Disease; Development Delay; Chromosome Abnormality; Hearing Loss; Dysmorphic Features; Skeletal Dysplasia; Congenital Abnormality; Microcephaly; Macrocephaly
MeSH Terms: conditions — Epilepsy; Neuromuscular Diseases; Intellectual Disability; Autism Spectrum Disorder; Muscle Hypotonia; Metabolism, Inborn Errors; Movement Disorders; Genetic Diseases, Inborn; Learning Disabilities; Chromosome Aberrations; Hearing Loss; Mucopolysaccharidosis IV; Congenital Abnormalities; Microcephaly; Megalencephaly

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The study coordinator will assign the first randomization to pre-visit preparation arm and care providers will not be told of the patient's pre-visit preparatory randomization arm prior to the first usual care visit. Randomization to exome sequencing will be performed after the first usual care visit by the study coordinator.
  Investigators will receive de-identified coded data and thus will not be able to link a patient name to an intervention arm. Some analyses will require individual-level randomization arm status to allow for comparison of parent questionnaire responses or health outcomes by arm - a major focus of this study.
  All interviewers and medical records staff conducting telephone surveys and/or medical records abstraction for clinical data will be blinded to the participants randomization status. Access to this information will be blocked in the electronic patient tracking status by study role.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Pre-visit prep / usual care + exome seq (Experimental): Participants randomized to pre-visit prep will receive a study packet with educational materials and a question prompt list. These participants will be instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to their clinic visit 1 appointment.
  Participants will receive usual care and will be offered research exome sequencing.
  Interventions: Behavioral: Pre-visit prep; Diagnostic Test: usual care + exome seq
- Pre-visit prep / usual care (Experimental): Participants randomized to pre-visit prep will receive a study packet with educational materials and a question prompt list. These participants will be instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to their clinic visit 1 appointment.
  Participants will receive usual care.
  Interventions: Behavioral: Pre-visit prep
- No prep / usual care + exome seq (Experimental): Participants in the no pre-visit preparation arm will receive a mailed card reminding them about their upcoming clinic visit.
  Participants will receive usual care and will be offered research exome sequencing.
  Interventions: Diagnostic Test: usual care + exome seq
- No prep / usual care (No Intervention): Participants in the no pre-visit preparation arm will receive a mailed card reminding them about their upcoming clinic visit.
  Participants will receive usual care.

INTERVENTIONS:
Behavioral: Pre-visit prep — Patient and provider surveys will be used to measure the impact of pre-visit preparation on the primary outcomes of engagement of participants in the clinical interaction and their view of the interaction as patient-centered, in addition to secondary outcomes that may be affected by this intervention (described above). The study investigators will test the hypothesis that patients will benefit from pre-visit preparation by: (1) rating their clinical encounters as more patient-centered and (2) asking more questions during their clinical encounters.
  Arms: Pre-visit prep / usual care; Pre-visit prep / usual care + exome seq
Diagnostic Test: usual care + exome seq — Provider surveys will be used to assess impact of exome sequencing on diagnostic thinking and management planning. Health utilization and condition-specific general clinical outcomes will be assessed from health records data.
  Arms: No prep / usual care + exome seq; Pre-visit prep / usual care + exome seq

SUMMARY:
The "North Carolina Clinical Genomic Evaluation by Next-gen Exome Sequencing, 2 (NCGENES 2)" study is part of a larger consortium project investigating the clinical utility, or net benefit of an intervention on patient and family well-being as well as diagnostic efficacy, management planning, and medical outcomes. A clinical trial will be implemented to compare (1) first-line exome sequencing to usual care and (2) participant pre-visit preparation to no pre-visit preparation. The study will use a randomized controlled design, with 2x2 factorial design, coupled with patient-reported outcomes and comprehensive clinical data collection addressing key outcomes, to determine the net impact of diagnostic results and secondary findings.

DETAILED DESCRIPTION:
The NCGENES 2 study is part of the "Clinical Sequencing Evidence-Generating Research (CSER2)" - Clinical Sites with Enhanced Diversity (U01), and brings together interdisciplinary experts from across North Carolina to address questions critical to the translation of genomic medicine to the care of patients with suspected genetic disorders.

In this renewal of the initial NCGENES study, NCGENES 2 will carry out a clinical trial of exome sequencing as a diagnostic test to answer the next set of questions vital to making genome-scale sequencing a routine clinical tool. The study population will be drawn from a state-wide network of Clinical Genetics and Pediatric Neurology clinics -- clinical domains in which patients are enriched for phenotypes caused by heterogeneous genetic conditions. Exome sequencing and genome sequencing (ES/GS) are efficient means of establishing a molecular diagnosis in these populations, with yields of positive or possible diagnostic results in at least 30% of patients examined based on findings from NCGENES and other work. Evidence will be generated regarding the clinical utility of ES/GS using a prospective randomized controlled trial that compares usual care plus exome sequencing to usual care. Patient-reported data, electronic health records data, and administrative claims data will be used to evaluate defined health outcomes, in collaboration with experts in health economics and health services research, to address pressing questions about the utility of exome sequencing. Furthermore, an examination of communication between patients and physicians, and between physicians and laboratories, and how these critical interactions affect the utility of genomic sequencing will be conducted. A second, nested randomized trial (crossed with exome sequencing in a full-factorial design) will be incorporated to test the hypothesis that a theory-based, multi-component pre-clinic preparation intervention for patients will improve patient-centered outcomes. An "embedded Ethical, Legal, and Social Implications (ELSI)" component will provide feedback to providers regarding communication discrepancies to iteratively improve care. Finally, the challenges of integrating clinical data and genomic information across a state-wide network of sites and examining different models of interaction between genomic clinicians and molecular diagnostic laboratorians will be explored.

ELIGIBILITY:
Both children and parents are participants:

Inclusion Criteria:

Parents meeting the following criteria:

1. Parent of a child who meets the criteria below
2. At least 18 years old.
3. Must be able to provide informed consent for child and self.
4. Must be fluent in English or Spanish.

Children meeting the following criteria:

1. Infants and children 15 years old or less.
2. Referred for initial evaluation of a possible monogenic disorder OR
3. Seen for evaluation of an undiagnosed disorder in a study-associated clinic.

Exclusion Criteria:

Parents:

1. Younger than 18 years old.
2. Unwilling to complete study surveys and other procedures.
3. Have cognitive or other impairments precluding ability to provide giving informed consent.
4. Not fluent in English or Spanish.
5. Unable to attend all clinic visits

Children:

1. Have a known genetic or non-genetic diagnosis (only referred for counseling or management).
2. Medically unstable.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2024-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette T Bensen, Ph.D, Study Director — University of North Carolina, Chapel Hill; Jonathan S Berg, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Mission Health, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with NIH mandates to share genetic data via submission of raw genotype calls from whole exome sequencing to the database of Genotypes and Phenotypes (dbGaP). All data that is submitted to dbGaP, including individual participant data, is anonymous and includes demographic variables: age of onset, birthplace, sex, race, education level, age. Data is uploaded in batches to the dbGaP website.
  Individual-level de-identified coded data will be available to investigators outside of the study team at the end of the study after publication of primary results. Investigators will apply for data by formal submission of a letter of intent that will be reviewed and approved by the study leadership. Investigators of approved projects will sign an inter-institution data sharing agreement (for investigators outside of the studies parent institution). The analytic data set will be shared with the investigator via a secure server restricted by password access.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared following study completion and publication of primary study results.
Access Criteria: Described above. Access will be by study leadership permission and under an inter-institutional data sharing agreement where relevant
URL: http://www.med.unc.edu/ncgenes

REFERENCES:
- [Background] Aboumatar HJ, Carson KA, Beach MC, Roter DL, Cooper LA. The impact of health literacy on desire for participation in healthcare, medical visit communication, and patient reported outcomes among patients with hypertension. J Gen Intern Med. 2013 Nov;28(11):1469-76. doi: 10.1007/s11606-013-2466-5. Epub 2013 May 21. PMID 23690237
- [Background] ACMG Board of Directors. Clinical utility of genetic and genomic services: a position statement of the American College of Medical Genetics and Genomics. Genet Med. 2015 Jun;17(6):505-7. doi: 10.1038/gim.2015.41. Epub 2015 Mar 12. PMID 25764213
- [Background] Amendola LM, Dorschner MO, Robertson PD, Salama JS, Hart R, Shirts BH, Murray ML, Tokita MJ, Gallego CJ, Kim DS, Bennett JT, Crosslin DR, Ranchalis J, Jones KL, Rosenthal EA, Jarvik ER, Itsara A, Turner EH, Herman DS, Schleit J, Burt A, Jamal SM, Abrudan JL, Johnson AD, Conlin LK, Dulik MC, Santani A, Metterville DR, Kelly M, Foreman AK, Lee K, Taylor KD, Guo X, Crooks K, Kiedrowski LA, Raffel LJ, Gordon O, Machini K, Desnick RJ, Biesecker LG, Lubitz SA, Mulchandani S, Cooper GM, Joffe S, Richards CS, Yang Y, Rotter JI, Rich SS, O'Donnell CJ, Berg JS, Spinner NB, Evans JP, Fullerton SM, Leppig KA, Bennett RL, Bird T, Sybert VP, Grady WM, Tabor HK, Kim JH, Bamshad MJ, Wilfond B, Motulsky AG, Scott CR, Pritchard CC, Walsh TD, Burke W, Raskind WH, Byers P, Hisama FM, Rehm H, Nickerson DA, Jarvik GP. Actionable exomic incidental findings in 6503 participants: challenges of variant classification. Genome Res. 2015 Mar;25(3):305-15. doi: 10.1101/gr.183483.114. Epub 2015 Jan 30. PMID 25637381
- [Background] Barnett ML, Landon BE, O'Malley AJ, Keating NL, Christakis NA. Mapping physician networks with self-reported and administrative data. Health Serv Res. 2011 Oct;46(5):1592-609. doi: 10.1111/j.1475-6773.2011.01262.x. Epub 2011 Apr 26. PMID 21521213
- [Background] Bates BR. Public culture and public understanding of genetics: a focus group study. Public Underst Sci. 2005 Jan;14(1):47-65. doi: 10.1177/0963662505048409. PMID 15822248
- [Background] Berg JS, Adams M, Nassar N, Bizon C, Lee K, Schmitt CP, Wilhelmsen KC, Evans JP. An informatics approach to analyzing the incidentalome. Genet Med. 2013 Jan;15(1):36-44. doi: 10.1038/gim.2012.112. Epub 2012 Sep 20. PMID 22995991
- [Background] Berg JS, Foreman AK, O'Daniel JM, Booker JK, Boshe L, Carey T, Crooks KR, Jensen BC, Juengst ET, Lee K, Nelson DK, Powell BC, Powell CM, Roche MI, Skrzynia C, Strande NT, Weck KE, Wilhelmsen KC, Evans JP. A semiquantitative metric for evaluating clinical actionability of incidental or secondary findings from genome-scale sequencing. Genet Med. 2016 May;18(5):467-75. doi: 10.1038/gim.2015.104. Epub 2015 Aug 13. PMID 26270767
- [Background] Black KZ, Hardy CY, De Marco M, Ammerman AS, Corbie-Smith G, Council B, Ellis D, Eng E, Harris B, Jackson M, Jean-Baptiste J, Kearney W, Legerton M, Parker D, Wynn M, Lightfoot A. Beyond incentives for involvement to compensation for consultants: increasing equity in CBPR approaches. Prog Community Health Partnersh. 2013 Fall;7(3):263-70. doi: 10.1353/cpr.2013.0040. PMID 24056508
- [Background] Brandes K, Linn AJ, Butow PN, van Weert JC. The characteristics and effectiveness of Question Prompt List interventions in oncology: a systematic review of the literature. Psychooncology. 2015 Mar;24(3):245-52. doi: 10.1002/pon.3637. Epub 2014 Jul 31. PMID 25082386
- [Background] Burkett K, Morris E, Manning-Courtney P, Anthony J, Shambley-Ebron D. African American families on autism diagnosis and treatment: the influence of culture. J Autism Dev Disord. 2015 Oct;45(10):3244-54. doi: 10.1007/s10803-015-2482-x. PMID 26055985
- [Background] Bussey-Jones J, Garrett J, Henderson G, Moloney M, Blumenthal C, Corbie-Smith G. The role of race and trust in tissue/blood donation for genetic research. Genet Med. 2010 Feb;12(2):116-21. doi: 10.1097/GIM.0b013e3181cd6689. PMID 20098329
- [Background] Catz DS, Green NS, Tobin JN, Lloyd-Puryear MA, Kyler P, Umemoto A, Cernoch J, Brown R, Wolman F. Attitudes about genetics in underserved, culturally diverse populations. Community Genet. 2005;8(3):161-72. doi: 10.1159/000086759. PMID 16113533
- [Background] Clayton JM, Butow PN, Tattersall MH, Devine RJ, Simpson JM, Aggarwal G, Clark KJ, Currow DC, Elliott LM, Lacey J, Lee PG, Noel MA. Randomized controlled trial of a prompt list to help advanced cancer patients and their caregivers to ask questions about prognosis and end-of-life care. J Clin Oncol. 2007 Feb 20;25(6):715-23. doi: 10.1200/JCO.2006.06.7827. PMID 17308275
- [Background] Corbie-Smith G, Thomas SB, St George DM. Distrust, race, and research. Arch Intern Med. 2002 Nov 25;162(21):2458-63. doi: 10.1001/archinte.162.21.2458. PMID 12437405
- [Background] Cunningham-Burley S. Public knowledge and public trust. Community Genet. 2006;9(3):204-10. doi: 10.1159/000092658. PMID 16741351
- [Background] DeWalt DA, Schillinger D, Ruo B, Bibbins-Domingo K, Baker DW, Holmes GM, Weinberger M, Macabasco-O'Connell A, Broucksou K, Hawk V, Grady KL, Erman B, Sueta CA, Chang PP, Cene CW, Wu JR, Jones CD, Pignone M. Multisite randomized trial of a single-session versus multisession literacy-sensitive self-care intervention for patients with heart failure. Circulation. 2012 Jun 12;125(23):2854-62. doi: 10.1161/CIRCULATIONAHA.111.081745. Epub 2012 May 9. PMID 22572916
- [Background] Dobransky-Fasiska D, Brown C, Pincus HA, Nowalk MP, Wieland M, Parker LS, Cruz M, McMurray ML, Mulsant B, Reynolds CF 3rd; RNDC-Community Partners. Developing a community-academic partnership to improve recognition and treatment of depression in underserved African American and white elders. Am J Geriatr Psychiatry. 2009 Nov;17(11):953-64. doi: 10.1097/JGP.0b013e31818f3a7e. PMID 20104053
- [Background] Durand MA, Carpenter L, Dolan H, Bravo P, Mann M, Bunn F, Elwyn G. Do interventions designed to support shared decision-making reduce health inequalities? A systematic review and meta-analysis. PLoS One. 2014 Apr 15;9(4):e94670. doi: 10.1371/journal.pone.0094670. eCollection 2014. PMID 24736389
- [Background] Eggly S, Harper FW, Penner LA, Gleason MJ, Foster T, Albrecht TL. Variation in question asking during cancer clinical interactions: a potential source of disparities in access to information. Patient Educ Couns. 2011 Jan;82(1):63-8. doi: 10.1016/j.pec.2010.04.008. Epub 2010 Apr 28. PMID 20430566
- [Background] Elder JH, Brasher S, Alexander B. Identifying the Barriers to Early Diagnosis and Treatment in Underserved Individuals with Autism Spectrum Disorders (ASD) and Their Families: A Qualitative Study. Issues Ment Health Nurs. 2016 Jun;37(6):412-20. doi: 10.3109/01612840.2016.1153174. Epub 2016 Apr 12. PMID 27070190
- [Background] Epstein RM, Street RL Jr. The values and value of patient-centered care. Ann Fam Med. 2011 Mar-Apr;9(2):100-3. doi: 10.1370/afm.1239. No abstract available. PMID 21403134
- [Background] Evans JP, Wilhelmsen KC, Berg J, Schmitt CP, Krishnamurthy A, Fecho K, Ahalt SC. A New Framework and Prototype Solution for Clinical Decision Support and Research in Genomics and Other Data-intensive Fields of Medicine. EGEMS (Wash DC). 2016 Apr 19;4(1):1198. doi: 10.13063/2327-9214.1198. eCollection 2016. PMID 27195307
- [Background] Evans JP. Return of results to the families of children in genomic sequencing: tallying risks and benefits. Genet Med. 2013 Jun;15(6):435-6. doi: 10.1038/gim.2013.54. No abstract available. PMID 23739673
- [Background] Evans JP. When is a medical finding "incidental"? Genet Med. 2013 Jul;15(7):515-6. doi: 10.1038/gim.2013.74. Epub 2013 May 30. No abstract available. PMID 23722872
- [Background] Facio FM, Lee K, O'Daniel JM. A genetic counselor's guide to using next-generation sequencing in clinical practice. J Genet Couns. 2014 Aug;23(4):455-62. doi: 10.1007/s10897-013-9662-7. Epub 2013 Oct 24. PMID 24151055
- [Background] Fan Z, Greenwood R, Felix AC, Shiloh-Malawsky Y, Tennison M, Roche M, Crooks K, Weck K, Wilhelmsen K, Berg J, Evans J. GCH1 heterozygous mutation identified by whole-exome sequencing as a treatable condition in a patient presenting with progressive spastic paraplegia. J Neurol. 2014 Mar;261(3):622-4. doi: 10.1007/s00415-014-7265-3. Epub 2014 Feb 8. No abstract available. PMID 24509643
- [Background] Foreman AK, Lee K, Evans JP. The NCGENES project: exploring the new world of genome sequencing. N C Med J. 2013 Nov-Dec;74(6):500-4. PMID 24316776
- [Background] Frey LJ, Lenert L, Lopez-Campos G. EHR Big Data Deep Phenotyping. Contribution of the IMIA Genomic Medicine Working Group. Yearb Med Inform. 2014 Aug 15;9(1):206-11. doi: 10.15265/IY-2014-0006. PMID 25123744
- [Background] Girdea M, Dumitriu S, Fiume M, Bowdin S, Boycott KM, Chenier S, Chitayat D, Faghfoury H, Meyn MS, Ray PN, So J, Stavropoulos DJ, Brudno M. PhenoTips: patient phenotyping software for clinical and research use. Hum Mutat. 2013 Aug;34(8):1057-65. doi: 10.1002/humu.22347. Epub 2013 May 24. PMID 23636887
- [Background] Gordon HS, Street RL Jr, Sharf BF, Souchek J. Racial differences in doctors' information-giving and patients' participation. Cancer. 2006 Sep 15;107(6):1313-20. doi: 10.1002/cncr.22122. PMID 16909424
- [Background] Gozu A, Beach MC, Price EG, Gary TL, Robinson K, Palacio A, Smarth C, Jenckes M, Feuerstein C, Bass EB, Powe NR, Cooper LA. Self-administered instruments to measure cultural competence of health professionals: a systematic review. Teach Learn Med. 2007 Spring;19(2):180-90. doi: 10.1080/10401330701333654. PMID 17564547
- [Background] Green RC, Berg JS, Grody WW, Kalia SS, Korf BR, Martin CL, McGuire AL, Nussbaum RL, O'Daniel JM, Ormond KE, Rehm HL, Watson MS, Williams MS, Biesecker LG; American College of Medical Genetics and Genomics. ACMG recommendations for reporting of incidental findings in clinical exome and genome sequencing. Genet Med. 2013 Jul;15(7):565-74. doi: 10.1038/gim.2013.73. Epub 2013 Jun 20. PMID 23788249
- [Background] Haase R, Michie M, Skinner D. Flexible positions, managed hopes: the promissory bioeconomy of a whole genome sequencing cancer study. Soc Sci Med. 2015 Apr;130:146-53. doi: 10.1016/j.socscimed.2015.02.016. Epub 2015 Feb 13. PMID 25697637
- [Background] Haga SB, Rosanbalm KD, Boles L, Tindall GM, Livingston TM, O'Daniel JM. Promoting public awareness and engagement in genome sciences. J Genet Couns. 2013 Aug;22(4):508-16. doi: 10.1007/s10897-013-9577-3. Epub 2013 Feb 23. PMID 23435715
- [Background] Hartz SM, Quan T, Ibiebele A, Fisher SL, Olfson E, Salyer P, Bierut LJ. The significant impact of education, poverty, and race on Internet-based research participant engagement. Genet Med. 2017 Feb;19(2):240-243. doi: 10.1038/gim.2016.91. Epub 2016 Jul 28. PMID 27467456
- [Background] Henderson GE. With great (participant) rights comes great (researcher) responsibility. Genet Med. 2016 Feb;18(2):124-5. doi: 10.1038/gim.2015.67. Epub 2015 May 7. No abstract available. PMID 25950735
- [Background] Hudon C, Fortin M, Haggerty JL, Lambert M, Poitras ME. Measuring patients' perceptions of patient-centered care: a systematic review of tools for family medicine. Ann Fam Med. 2011 Mar-Apr;9(2):155-64. doi: 10.1370/afm.1226. PMID 21403143
- [Background] Isaacson M. Clarifying concepts: cultural humility or competency. J Prof Nurs. 2014 May-Jun;30(3):251-8. doi: 10.1016/j.profnurs.2013.09.011. PMID 24939335
- [Background] Joseph-Williams N, Elwyn G, Edwards A. Knowledge is not power for patients: a systematic review and thematic synthesis of patient-reported barriers and facilitators to shared decision making. Patient Educ Couns. 2014 Mar;94(3):291-309. doi: 10.1016/j.pec.2013.10.031. Epub 2013 Nov 9. PMID 24305642
- [Background] Kaphingst KA, Blanchard M, Milam L, Pokharel M, Elrick A, Goodman MS. Relationships Between Health Literacy and Genomics-Related Knowledge, Self-Efficacy, Perceived Importance, and Communication in a Medically Underserved Population. J Health Commun. 2016;21 Suppl 1(Suppl 1):58-68. doi: 10.1080/10810730.2016.1144661. PMID 27043759
- [Background] Katz MG, Jacobson TA, Veledar E, Kripalani S. Patient literacy and question-asking behavior during the medical encounter: a mixed-methods analysis. J Gen Intern Med. 2007 Jun;22(6):782-6. doi: 10.1007/s11606-007-0184-6. Epub 2007 Apr 12. PMID 17431697
- [Background] Kinnersley P, Edwards A, Hood K, Ryan R, Prout H, Cadbury N, MacBeth F, Butow P, Butler C. Interventions before consultations to help patients address their information needs by encouraging question asking: systematic review. BMJ. 2008 Jul 16;337:a485. doi: 10.1136/bmj.a485. PMID 18632672
- [Background] Lea DH, Kaphingst KA, Bowen D, Lipkus I, Hadley DW. Communicating genetic and genomic information: health literacy and numeracy considerations. Public Health Genomics. 2011;14(4-5):279-89. doi: 10.1159/000294191. Epub 2010 Apr 20. PMID 20407217
- [Background] Lee K, Berg JS, Milko L, Crooks K, Lu M, Bizon C, Owen P, Wilhelmsen KC, Weck KE, Evans JP, Garg S. High Diagnostic Yield of Whole Exome Sequencing in Participants With Retinal Dystrophies in a Clinical Ophthalmology Setting. Am J Ophthalmol. 2015 Aug;160(2):354-363.e9. doi: 10.1016/j.ajo.2015.04.026. Epub 2015 Apr 22. PMID 25910913
- [Background] Leos C, Khan CM, Rini C. Understanding self-management behaviors in symptomatic adults with uncertain etiology using an illness perceptions framework. J Behav Med. 2016 Apr;39(2):310-9. doi: 10.1007/s10865-015-9698-2. Epub 2015 Dec 8. PMID 26646840
- [Background] Nutter RL, Bullas LR, Schultz RL. Some properties of five new Salmonella bacteriophages. J Virol. 1970 Jun;5(6):754-64. doi: 10.1128/JVI.5.6.754-764.1970. PMID 4193833
- [Background] O'Daniel JM, Lee K. Whole-genome and whole-exome sequencing in hereditary cancer: impact on genetic testing and counseling. Cancer J. 2012 Jul-Aug;18(4):287-92. doi: 10.1097/PPO.0b013e318262467e. PMID 22846728
- [Background] O'Daniel JM, Rosanbalm KD, Boles L, Tindall GM, Livingston TM, Haga SB. Enhancing geneticists' perspectives of the public through community engagement. Genet Med. 2012 Feb;14(2):243-9. doi: 10.1038/gim.2011.29. Epub 2012 Jan 19. PMID 22241095
- [Background] Pickard KE, Kilgore AN, Ingersoll BR. Using Community Partnerships to Better Understand the Barriers to Using an Evidence-Based, Parent-Mediated Intervention for Autism Spectrum Disorder in a Medicaid System. Am J Community Psychol. 2016 Jun;57(3-4):391-403. doi: 10.1002/ajcp.12050. Epub 2016 May 19. PMID 27216766
- [Background] Roche MI, Berg JS. Incidental Findings with Genomic Testing: Implications for Genetic Counseling Practice. Curr Genet Med Rep. 2015;3(4):166-176. doi: 10.1007/s40142-015-0075-9. Epub 2015 Aug 25. PMID 26566463
- [Background] Rodriguez V, Andrade AD, Garcia-Retamero R, Anam R, Rodriguez R, Lisigurski M, Sharit J, Ruiz JG. Health literacy, numeracy, and graphical literacy among veterans in primary care and their effect on shared decision making and trust in physicians. J Health Commun. 2013;18 Suppl 1(Suppl 1):273-89. doi: 10.1080/10810730.2013.829137. PMID 24093361
- [Background] Sansoni JE, Grootemaat P, Duncan C. Question Prompt Lists in health consultations: A review. Patient Educ Couns. 2015 Jun 3:S0738-3991(15)00258-X. doi: 10.1016/j.pec.2015.05.015. Online ahead of print. PMID 26104993
- [Background] Sawaya GF, Guirguis-Blake J, LeFevre M, Harris R, Petitti D; U.S. Preventive Services Task Force. Update on the methods of the U.S. Preventive Services Task Force: estimating certainty and magnitude of net benefit. Ann Intern Med. 2007 Dec 18;147(12):871-5. doi: 10.7326/0003-4819-147-12-200712180-00007. PMID 18087058
- [Background] Say R, Murtagh M, Thomson R. Patients' preference for involvement in medical decision making: a narrative review. Patient Educ Couns. 2006 Feb;60(2):102-14. doi: 10.1016/j.pec.2005.02.003. PMID 16442453
- [Background] Seifert BA, O'Daniel JM, Amin K, Marchuk DS, Patel NM, Parker JS, Hoyle AP, Mose LE, Marron A, Hayward MC, Bizon C, Wilhelmsen KC, Evans JP, Earp HS 3rd, Sharpless NE, Hayes DN, Berg JS. Germline Analysis from Tumor-Germline Sequencing Dyads to Identify Clinically Actionable Secondary Findings. Clin Cancer Res. 2016 Aug 15;22(16):4087-4094. doi: 10.1158/1078-0432.CCR-16-0015. Epub 2016 Apr 15. PMID 27083775
- [Background] Skrzynia C, Berg JS, Willis MS, Jensen BC. Genetics and heart failure: a concise guide for the clinician. Curr Cardiol Rev. 2015;11(1):10-7. doi: 10.2174/1573403x09666131117170446. PMID 24251456
- [Background] Strande NT, Berg JS. Defining the Clinical Value of a Genomic Diagnosis in the Era of Next-Generation Sequencing. Annu Rev Genomics Hum Genet. 2016 Aug 31;17:303-32. doi: 10.1146/annurev-genom-083115-022348. Epub 2016 May 26. PMID 27362341
- [Background] van Nimwegen KJ, Schieving JH, Willemsen MA, Veltman JA, van der Burg S, van der Wilt GJ, Grutters JP. The diagnostic pathway in complex paediatric neurology: a cost analysis. Eur J Paediatr Neurol. 2015 Mar;19(2):233-9. doi: 10.1016/j.ejpn.2014.12.014. Epub 2014 Dec 29. PMID 25604808
- [Background] Willems S, De Maesschalck S, Deveugele M, Derese A, De Maeseneer J. Socio-economic status of the patient and doctor-patient communication: does it make a difference? Patient Educ Couns. 2005 Feb;56(2):139-46. doi: 10.1016/j.pec.2004.02.011. PMID 15653242
- [Background] Zamora I, Williams ME, Higareda M, Wheeler BY, Levitt P. Brief Report: Recruitment and Retention of Minority Children for Autism Research. J Autism Dev Disord. 2016 Feb;46(2):698-703. doi: 10.1007/s10803-015-2603-6. PMID 26404703
- [Derived] Staley BS, Milko LV, Waltz M, Griesemer I, Mollison L, Grant TL, Farnan L, Roche M, Navas A, Lightfoot A, Foreman AKM, O'Daniel JM, O'Neill SC, Lin FC, Roman TS, Brandt A, Powell BC, Rini C, Berg JS, Bensen JT. Evaluating the clinical utility of early exome sequencing in diverse pediatric outpatient populations in the North Carolina Clinical Genomic Evaluation of Next-generation Exome Sequencing (NCGENES) 2 study: a randomized controlled trial. Trials. 2021 Jun 14;22(1):395. doi: 10.1186/s13063-021-05341-2. PMID 34127041
- See also: Ales M, Luca L, Marija V, Gorazd R, Karin W, Ana B, Alenka H, Peterlin B. Phenotype-driven gene target definition in clinical genome-wide sequencing data interpretation. Genet Med [Internet]. 2016 Mar 31 [cited 2016 Aug 3] — http://www.nature.com/gim/journal/vaop/ncurrent/full/gim201622a.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 927 children were eligible for recruitment, and of these 791 parents/caregivers were approached by phone prior to their clinic visit; 514 parents/caregivers were reached for a recruitment phone call, and a total of 417 dyads consisting of a child and their parent/caregiver were enrolled and consented to randomization. Of these, 274 baseline intake forms were obtained at a clinic visit and those dyads continued in the study, for a total of 548 individuals enrolled in the protocol.
Groups:
- Parent/Caregiver Pre-visit Prep + Exome; Child Pre-visit Prep + Exome: Dyads (parent/caregiver + child) that are randomized to the "pre-visit prep" arm receive a study packet with educational materials and a question prompt list. The parent/caregiver is instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to the child's clinic visit 1 appointment.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads that are randomized to the "exome" arm are offered exome sequencing in addition to tests ordered by the physician at that visit. The parent/caregiver may decline for their child to have exome sequencing at this point.
- Parent/Caregiver Pre-visit Prep + Usual Care; Child Pre-visit Prep + Usual Care: Dyads (parent/caregiver + child) that are randomized to the "pre-visit prep" arm receive a study packet with educational materials and a question prompt list. The parent/caregiver is instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to the child's clinic visit 1 appointment.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads that are randomized to the "usual care" arm are not offered additional exome sequencing.
- Parent/Caregiver No Pre-visit Prep + Exome; Child No Pre-visit Prep + Exome: Dyads (parent/caregiver + child) that are randomized to the "no pre-visit prep" arm receive a mailed card reminding them about their upcoming clinic visit.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads that are randomized to the "exome" arm are offered exome sequencing in addition to tests ordered by the physician at that visit. The parent/caregiver may decline for their child to have exome sequencing at this point.
- Parent/Caregiver No Pre-visit Prep + Usual Care; Child No Pre-visit Prep + Usual Care: Dyads (parent/caregiver + child) that are randomized to the "no pre-visit prep" arm receive a mailed card reminding them about their upcoming clinic visit.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads that are randomized to the "usual care" arm are not offered additional exome sequencing.
Period: Clinical Study
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Started (A total of 274 dyads (parent/caregiver + child) entered the protocol after being randomized in a 4 factorial design.) | 64 | 72 | 63 | 75 | 64 | 72 | 63 | 75
Second Stage Randomization and Consent Discussion (The 274 dyads who completed the clinic visit underwent a secondary consent discussion for randomization of the child participant to exome sequencing or usual care. Of these, 250 agreed to be randomized. Only the child participant was involved in this aspect of the study.) | 0 (Parent/caregiver participants were not involved in the Exome portion of the study.) | 0 (Parent/caregiver participants were not involved in the Exome portion of the study.) | 0 (Parent/caregiver participants were not involved in the Exome portion of the study.) | 0 (Parent/caregiver participants were not involved in the Exome portion of the study.) | 53 | 70 | 59 | 68
Completed | 64 | 72 | 63 | 75 | 53 | 70 | 59 | 68
Not Completed | 0 | 0 | 0 | 0 | 11 | 2 | 4 | 7
Period: Health Care Records Analysis
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Started (Health care records analyses were conducted for child participants who completed the clinical study.) | 0 (Parent/caregiver participants were not part of the health care records analysis portion of the study.) | 0 (Parent/caregiver participants were not part of the health care records analysis portion of the study.) | 0 (Parent/caregiver participants were not part of the health care records analysis portion of the study.) | 0 (Parent/caregiver participants were not part of the health care records analysis portion of the study.) | 53 | 70 | 59 | 68
6 Month Data Pre and Post (These numbers reflect the child participants in each of the four subgroups for whom 6-months of EHR data pre- and post- return of results were available to study.) | 0 | 0 | 0 | 0 | 26 | 36 | 32 | 38
Completed (These numbers reflect the child participants in each of the four subgroups for whom a complete set of EHR data (12 months pre- and post- return of results) were available.) | 0 | 0 | 0 | 0 | 22 | 35 | 27 | 31
Not Completed | 0 | 0 | 0 | 0 | 31 | 35 | 32 | 37

BASELINE CHARACTERISTICS:
Population: 274 dyads were randomized to the four study groups
Groups:
- Parent/Caregiver Pre-visit Prep + Exome; Child Pre-visit Prep + Exome: Dyads (parent/caregiver + child) randomized to the "pre-visit prep" arm receive a study packet with educational materials and a question prompt list. The parent/caregiver is instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to the child's clinic visit 1 appointment.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads randomized to the "exome" arm are offered exome sequencing in addition to tests ordered by the physician at that visit. The parent/caregiver may decline for their child to have exome sequencing at this point.
- Parent/Caregiver Pre-visit Prep + Usual Care; Child Pre-visit Prep + Usual Care: Dyads (parent/caregiver + child) randomized to the "pre-visit prep" arm receive a study packet with educational materials and a question prompt list. The parent/caregiver is instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to the child's clinic visit 1 appointment.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads randomized to the "usual care" arm are not offered additional exome sequencing.
- Parent/Caregiver No Pre-visit Prep + Exome; Child No Pre-visit Prep + Exome: Dyads (parent/caregiver + child) randomized to the "no pre-visit prep" arm receive a mailed card reminding them about their upcoming clinic visit.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads randomized to the "exome" arm are offered exome sequencing in addition to tests ordered by the physician at that visit. The parent/caregiver may decline for their child to have exome sequencing at this point.
- Parent/Caregiver No Pre-visit Prep + Usual Care; Child No Pre-visit Prep + Usual Care: Dyads (parent/caregiver + child) randomized to the "no pre-visit prep" arm receive a mailed card reminding them about their upcoming clinic visit.
  During the clinic visit 1 evaluation, the physician orders any tests deemed clinically appropriate. After completing the clinic visit, dyads randomized to the "usual care" arm are not offered additional exome sequencing.
- Total: Total of all reporting groups
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care | Total
Number analyzed (Participants) | 64 | 72 | 63 | 75 | 64 | 72 | 63 | 75 | 548
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (6.7) | 35.8 (7.0) | 36.6 (9.5) | 35.3 (9.3) | 5.4 (4.3) | 5.1 (4.3) | 6.8 (4.6) | 6.2 (4.1) | 20.8 (16.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 59 | 67 | 58 | 67 | 28 | 31 | 24 | 37 | 371
  Male | 3 | 3 | 4 | 6 | 36 | 41 | 39 | 38 | 170
  Did not answer | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could select any number of categories that represented their race/ethnicity. Therefore, the summed numbers may exceed the number of participants.
  Participants
    American Indian, Native American, or Alaska Native | 2 | 4 | 3 | 4 | 1 | 4 | 3 | 2 | 23
    Asian | 0 | 2 | 0 | 2 | 3 | 2 | 1 | 3 | 13
    Black or African American | 7 | 11 | 10 | 5 | 8 | 14 | 10 | 7 | 72
    Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White or European American | 52 | 49 | 49 | 54 | 49 | 50 | 48 | 57 | 408
    Middle Eastern or North African/Mediterranean | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
    Hispanic/Latino(a) | 4 | 5 | 2 | 10 | 7 | 7 | 2 | 13 | 50
    Prefer not to answer | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
    Unknown/none of these fully describe me | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Initial Patient Pediatric Quality of Life (Peds QL) Score
Description: The Peds QL Measurement Model for the Pediatric Quality of Inventory measures the core dimensions of health as delineated by the World Health Organization as well as role (school) functioning. The 23-item PedsQL Core Scales (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning) are developmentally appropriate surveys (Ages 2-4, 5-7, 8-12, 13-18) designed for parent proxy report. The 23 items are grouped together on the questionnaire, and are answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better Health-Related Quality of Life (HRQOL). This questionnaire will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 62 | 70 | 61 | 72
score on a scale | 64.37 (20.59) | 65.83 (18.00) | 60.04 (17.10) | 63.39 (18.49)

2. Primary Outcome: Final Patient Pediatric Quality of Life (Peds QL) Score
Description: The Peds QL Measurement Model for the Pediatric Quality of Inventory measures the core dimensions of health as delineated by the World Health Organization as well as role (school) functioning. The 23-item PedsQL Core Scales (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning) are developmentally appropriate surveys (Ages 2-4, 5-7, 8-12, 13-18) designed for parent proxy report. The 23 items are grouped together on the questionnaire, and are answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better HRQOL. This questionnaire will be interviewer administered by telephone.
Time Frame: 6 months after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 36 | 26 | 30
score on a scale | 72.15 (17.95) | 75.74 (15.01) | 71.65 (17.10) | 68.90 (19.01)

3. Primary Outcome: Initial Caregiver QoL Score
Description: The Short-Form Health Survey (SF-12) questionnaire is a reliable measure of perceived health that describes the degree of general physical health status and mental health distress. It consists of 12 items, derived from the physical and mental domains. Scores have a range of 0 to 100 and were designed to have a mean score of 50 and a standard deviation of 10 in a representative sample of the US population, with higher scores indicating greater functioning. This questionnaire will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 50 | 55 | 48 | 55
score on a scale | 50.14 (10.25) | 48.84 (8.14) | 51.30 (8.72) | 47.69 (9.59)

4. Primary Outcome: Intermediate Caregiver QoL Score
Description: The SF-12 questionnaire is a reliable measure of perceived health that describes the degree of general physical health status and mental health distress. It consists of 12 items, derived from the physical and mental domains. Scores have a range of 0 to 100 and were designed to have a mean score of 50 and a standard deviation of 10 in a representative sample of the US population, with higher scores indicating greater functioning. This questionnaire will be interviewer administered by telephone.
Time Frame: 2 weeks after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 19 | 28 | 24 | 31
score on a scale | 51.48 (9.03) | 46.58 (9.68) | 50.66 (11.49) | 50.08 (7.52)

5. Primary Outcome: Final Caregiver QoL Score
Description: as for outcome 4
Time Frame: 6 months after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 38 | 26 | 30
score on a scale | 53.31 (5.41) | 50.38 (8.21) | 47.41 (11.44) | 47.46 (10.39)

6. Primary Outcome: Post-Clinic Visit 1 Mean Patient Centeredness Score
Description: Patient centeredness scale, which measures the caregiver's perception of the level of patient centeredness of their visit with their child's provider (developed by Little et al., 2001). Self-administered in the clinic, immediately after clinic visit 1. Item responses will be coded as: 1=Very strongly disagree; 2=Strongly disagree; 3=Moderately disagree; 4=Neither agree nor disagree; 5=Moderately agree; 6=Strongly agree; 7=Very strongly agree. Response values will be summed and divided by the total number of items (21) to obtain mean scores ranging from 0-7 where higher values indicate stronger perceptions of patient centeredness.
Time Frame: Immediately after clinic 1 day of visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 49 | 56 | 51 | 58
score on a scale | 5.7 (0.8) | 5.7 (0.9) | 5.9 (0.7) | 5.8 (0.9)

7. Primary Outcome: Post-Return of Results Mean Patient Centeredness Score
Description: as for outcome 6
Time Frame: 2 weeks after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 24 | 24 | 22
score on a scale | 5.5 (0.9) | 5 (1.3) | 5 (1.1) | 4.8 (1.6)

8. Primary Outcome: Number of Questions Caregiver Asks in Clinic Visit 1
Description: Count of number of questions caregiver asks provider in the audio recording of clinic visit 1. Coded by trained study staff.
Time Frame: During clinic 1 day of visit 1
Population: This analysis is conducted among the parent/caregiver participants who attended a clinic visit that was transcribed (a subset of all dyads who completed Clinic Visit 1). The analysis populations only represent the first randomization (Pre-visit prep vs. No pre-visit prep) because the second randomization (Exome vs. Usual care) did not occur until after the clinic visit was completed, and was therefore not germane to this specific outcome measure.
Measure: Mean (Standard Deviation); unit: Number of questions asked
Groups:
- Parent/Caregiver Pre-visit Prep: Dyads (parent/caregiver + child) that are randomized to the "pre-visit prep" arm receive a study packet with educational materials and a question prompt list. The parent/caregiver is instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to the child's clinic visit 1 appointment.
- Parent/Caregiver No Pre-visit Prep: Dyads (parent/caregiver + child) that are randomized to the "no pre-visit prep" arm receive a mailed card reminding them about their upcoming clinic visit.
Arm/Group | Parent/Caregiver Pre-visit Prep | Parent/Caregiver No Pre-visit Prep
Number analyzed (Participants) | 59 | 53
Number of questions asked | 4.36 (4.66) | 2.83 (3.03)

9. Primary Outcome: Number of In-patient Hospital Admissions Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of in-patient hospital admissions among child participants during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Admissions were summed across all participants.
Time Frame: 1 year prior to return of results
Population: This analysis includes the subset of child participants with 12 months of EHR data available before and after study results were returned.
Measure: Number; unit: In-patient hospital admissions
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
In-patient hospital admissions | 0 | 3 | 4 | 2

10. Primary Outcome: Number of In-patient Hospital Admissions Among Child Participants 1 Year After Return of Results
Description: Count of number of in-patient hospital admissions among child participants during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Admissions were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: In-patient hospital admissions
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
In-patient hospital admissions | 1 | 1 | 8 | 2

11. Primary Outcome: Number of In-patient Hospital Days Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of in-patient hospital days among child participants during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Days were summed across all participants.
Time Frame: 1 year prior to return of results
Population: as for outcome 9
Measure: Number; unit: In-patient hospital days
Groups:
- Pre-visit Prep + Exome: Participants randomized to pre-visit prep will receive a study packet with educational materials and a question prompt list. These participants will be instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to their clinic visit 1 appointment.
  After completing the clinic visit, participants are randomized to be offered exome sequencing in addition to the usual care they receive as part of their clinical evaluation. Parents may decline for their child to have exome sequencing at this point.
- Pre-visit Prep + Usual Care: Participants randomized to pre-visit prep will receive a study packet with educational materials and a question prompt list. These participants will be instructed to review the materials, discuss them with family members if desired, use the question prompt list to select questions they would like to ask at clinic visit 1, and bring the list to their clinic visit 1 appointment.
  After completing the clinic visit, participants are randomized to receive usual care as part of their clinical evaluation.
- No Pre-visit Prep + Exome: Participants randomized to the no pre-visit preparation arm will receive a mailed card reminding them about their upcoming clinic visit.
  After completing the clinic visit, participants are randomized to be offered exome sequencing in addition to the usual care they receive as part of their clinical evaluation. Parents may decline for their child to have exome sequencing at this point.
- No Pre-visit Prep + Usual Care: Participants randomized to the no pre-visit preparation arm will receive a mailed card reminding them about their upcoming clinic visit.
  After completing the clinic visit, participants are randomized to receive usual care as part of their clinical evaluation.
Arm/Group | Pre-visit Prep + Exome | Pre-visit Prep + Usual Care | No Pre-visit Prep + Exome | No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
In-patient hospital days | 0 | 13 | 22 | 1

12. Primary Outcome: Number of In-patient Hospital Days Among Child Participants 1 Year After Return of Results
Description: Count of number of in-patient hospital days among child participants during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Days were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: In-patient hospital days
Arm/Group | Pre-visit Prep + Exome | Pre-visit Prep + Usual Care | No Pre-visit Prep + Exome | No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
In-patient hospital days | 5 | 5 | 148 | 11

13. Primary Outcome: Number of Long-term Care Admissions Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of long-term care admissions among child participants during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Admissions were summed across all participants.
Time Frame: 1 year prior to return of results
Population: as for outcome 9
Measure: Number; unit: Long-term care admissions
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Long-term care admissions | 0 | 0 | 4 | 0

14. Primary Outcome: Number of Long-term Care Admissions Among Child Participants 1 Year After Return of Results
Description: Count of number of long-term care admissions among child participants during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Admissions were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: Long-term care admissions
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Long-term care admissions | 0 | 0 | 3 | 0

15. Primary Outcome: Number of Long-term Care Days Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of long-term care days among child participants during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Days were summed across all participants.
Time Frame: 1 year prior to return of results
Population: as for outcome 9
Measure: Number; unit: Long-term care days
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Long-term care days | 0 | 0 | 29 | 0

16. Primary Outcome: Number of Long-term Care Days Among Child Participants 1 Year After Return of Results
Description: Count of number of long-term care days during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Days were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: Long-term care days
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Long-term care days | 0 | 0 | 17 | 0

17. Primary Outcome: Number of ER Visits Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of ER visits during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Visits were summed across all participants.
Time Frame: 1 year prior to return of results
Population: as for outcome 9
Measure: Number; unit: ER visits
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
ER visits | 15 | 25 | 35 | 35

18. Primary Outcome: Number of ER Visits Among Child Participants 1 Year After Return of Results
Description: Count of number of ER visits during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Visits were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: ER visits
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
ER visits | 10 | 29 | 20 | 23

19. Primary Outcome: Number of Specialists Visits Among Child Participants 1 Year Prior to Return of Results
Description: Count of number of specialists visits during 1 year prior to return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Visits were summed across all participants.
Time Frame: 1 year prior to return of results
Population: as for outcome 9
Measure: Number; unit: Specialist visits
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Specialist visits | 202 | 665 | 663 | 332

20. Primary Outcome: Number of Specialists Visits Among Child Participants 1 Year After Return of Results
Description: Count of number of specialists visits during 1 year after return of results using data obtained from the Electronic Medical Record. Coded by trained study staff. Visits were summed across all participants.
Time Frame: 1 year after return of results
Population: as for outcome 9
Measure: Number; unit: Specialist visits
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 22 | 35 | 27 | 31
Specialist visits | 220 | 556 | 650 | 273

21. Secondary Outcome: Initial Average Peds QL Score for "Missing School for Not Feeling Well"
Description: This is a single item measure from the Peds QL that will be answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better HRQOL for this single measure. This questionnaire will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only. The parent/caregiver completes this measure as a proxy for the child.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 36 | 40 | 42 | 50
score on a scale | 70.8 (29.8) | 80.6 (20.5) | 65.5 (28.3) | 73 (28.7)

22. Secondary Outcome: Final Average Peds QL Score for "Missing School for Not Feeling Well"
Description: This is a single item measure from the Peds QL that will be answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better HRQOL for this single measure. This questionnaire will be interviewer-administered by telephone.
Time Frame: 6 months after return of results
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 12 | 23 | 19 | 20
score on a scale | 77.1 (23.8) | 82.6 (22.6) | 78.9 (23.3) | 81.3 (22.2)

23. Secondary Outcome: Initial Average Peds QL Score for "Missing School for Doctors Visit"
Description: This is a single item measure from the Peds QL that will be answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better HRQOL for this single measure. This measure will be included in the questionnaire that will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 36 | 40 | 41 | 50
score on a scale | 59.7 (28.4) | 65 (27.8) | 54.9 (27.2) | 60 (26.9)

24. Secondary Outcome: Final Average Peds QL Score for "Missing School for Doctors Visit"
Description: This is a single item measure from the Peds QL that will be answered on a scale of 0-4. Items are reversed scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better HRQOL for this single measure. This measure will be interviewer administered by telephone.
Time Frame: 6 months after return of results
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 12 | 23 | 19 | 20
score on a scale | 77.1 (23.8) | 82.6 (21.4) | 78.9 (23.3) | 82.5 (19.5)

25. Secondary Outcome: Initial Amount of Work Missed Because of Child's Condition or Treatments Score
Description: This is a single item measure that will be answered on a scale of 1-6 where 1=None, 2=Less than a week, 3=Between 1 and 4 weeks, 4= Between 4 and 8 weeks, 5=Between 8 and 12 weeks, 6=I stopped working altogether. Higher scores indicate greater amounts of work missed because of the child's condition or treatments. This measure will be included in the questionnaire that will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 62 | 70 | 61 | 72
score on a scale | 2.3 (1.7) | 2.4 (1.9) | 2.5 (1.8) | 2 (1.4)

26. Secondary Outcome: Final Amount of Work Missed Because of Child's Condition or Treatments Score
Description: This is a single item measure that will be answered on a scale of 1-6 where 1=None, 2=Less than a week, 3=Between 1 and 4 weeks, 4= Between 4 and 8 weeks, 5=Between 8 and 12 weeks, 6=I stopped working altogether. Higher scores indicate greater amounts of work missed because of the child's condition or treatments. This measure will be interviewer-administered by telephone.
Time Frame: 6 months after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 38 | 26 | 28
score on a scale | 2.3 (1.7) | 2.3 (1.8) | 2.5 (1.8) | 2.6 (2)

27. Secondary Outcome: Initial Difficulty With Finishing Normal Work (Including Both Work Outside of the Home and Housework) Because of Child's Condition or Treatments Score
Description: This is a single item measure that will be answered on a scale of 1-5, where 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. Higher scores indicate greater difficulty finishing normal work (including both work outside of the home and housework) because of child's condition or treatments. This measure will be included in the questionnaire that will be self-administered at home.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 62 | 70 | 62 | 72
score on a scale | 2.7 (1.4) | 2.5 (1.3) | 2.7 (1.2) | 2.4 (1.2)

28. Secondary Outcome: Intermediate Difficulty With Finishing Normal Work (Including Both Work Outside of the Home and Housework) Because of Child's Condition or Treatments Score
Description: This is a single item measure that will be answered on a scale of 1-5, where 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. Higher scores indicate greater difficulty finishing normal work (including both work outside of the home and housework) because of child's condition or treatments. This measure will be interviewer-administered by telephone.
Time Frame: 2 weeks after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 28 | 23 | 31
score on a scale | 1.9 (1.1) | 2 (1.1) | 2.3 (1.3) | 2.1 (1.1)

29. Secondary Outcome: Final Difficulty With Finishing Normal Work (Including Both Work Outside of the Home and Housework) Because of Child's Condition or Treatments Score
Description: as for outcome 28
Time Frame: 6 months after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 38 | 26 | 28
score on a scale | 2.1 (1.4) | 2.1 (1.3) | 2.1 (1.1) | 2.1 (1.2)

30. Secondary Outcome: Percent Concordance of Caregiver and Provider Reports of Genetic or Genomic Test Results
Description: Concordance between caregiver and provider reports of whether patients' diagnostic results were positive, negative, or uncertain. Coded as a dichotomous variable: 0=discordant diagnostic reports; 1=concordant diagnostic reports. Results are given as the number of parent/caregiver participant responses for each group that were concordant with the provider's diagnostic interpretation of the exome results.
Time Frame: 2 weeks after return of results
Population: This analysis is only performed in the subset of parent/caregiver participants whose child was randomized to receive exome sequencing and received an interpretation of their exome data from a provider.
Measure: Number; unit: participants
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Exome
Number analyzed (Participants) | 11 | 18
participants | 9 | 12

31. Secondary Outcome: Mean Baseline Self Efficacy Score
Description: Self-efficacy scale, which measures caregivers' confidence in communicating with their child's provider. Self-administered as part of the intake questionnaire. Measured with adapted Decision Self Efficacy Scale (developed by O'Connor, 1995). Adapted wording from the original scale so items refer to general communication, as opposed to a specific decision. Shorted scale to 7 items from 11 since not all items were applicable to this study. Item responses will be coded as: 1=Not at all confident; 5=Very confident. Mean scores will be calculated by summing the response values and dividing by the total number of items (7). Higher scores indicate higher confidence in communicating with their child's provider.
Time Frame: 4-6 weeks prior to clinic visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 72 | 70 | 62 | 73
score on a scale | 4.5 (0.5) | 4.5 (0.6) | 4.6 (0.4) | 4.6 (0.5)

32. Secondary Outcome: Mean Pre-Clinic Visit 1 Self Efficacy Score
Description: as for outcome 31
Time Frame: Immediately before Clinic Visit 1
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 28 | 24 | 31
score on a scale | 4.6 (0.5) | 4.4 (0.8) | 4.5 (0.5) | 4.4 (0.6)

33. Secondary Outcome: Post-Return of Results Mean FACToR Uncertainty Subscale Score
Description: Subscale of the Feeling About genomiC Testing Results measure assesses caregivers' level of uncertainty about their child's genetic test results (developed by Gallego et al., 2014). Interviewer administered by telephone. Item responses will be coded as: 1=Not at all; 2=A little; 3=Somewhat; 4=A good deal; 5=A great deal. Mean scores will be calculated by summing the response values and dividing by the total number of items (3). Higher scores indicate greater uncertainty about their child's genetic test results.
Time Frame: 2 weeks after return of results
Population: This analysis is conducted among the parent/caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent/Caregiver Pre-visit Prep + Exome | Parent/Caregiver Pre-visit Prep + Usual Care | Parent/Caregiver No Pre-visit Prep + Exome | Parent/Caregiver No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 20 | 24 | 23 | 21
score on a scale | 1.7 (0.6) | 2.4 (1.1) | 2.3 (1) | 2.2 (1.1)

34. Secondary Outcome: Vital Status at Final f/u
Description: Based on NC Vital Statistics, the child's vital status will be reported as living or deceased.
Time Frame: Final follow-up, up to approximately three years after clinic visit 1
Population: Child participants for whom sufficient data was available to determine vital status at follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 28 | 39 | 35 | 36
Participants
  Living | 28 | 38 | 35 | 36
  Deceased | 0 | 1 | 0 | 0

35. Secondary Outcome: Number of Child Participants With Causes of Death Unrelated to the Study
Description: Child causes of death related to the primary condition based on NC Vital Statistics, child causes of death will be reported as related to the disorder of the child or not related to the disorder of the child.
Time Frame: Final follow-up, up to approximately three years after clinic visit 1
Population: One child participant died during the course of the study follow-up period, unrelated to the study intervention. Cause of death was multiple organ failure and septic shock.
Measure: Count of Participants; unit: Participants
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
Number analyzed (Participants) | 0 | 1 | 0 | 0
Participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Child Pre-visit Prep + Exome | Child Pre-visit Prep + Usual Care | Child No Pre-visit Prep + Exome | Child No Pre-visit Prep + Usual Care
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/70 | 0/59 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/70 | 0/59 | 0/68
Other Adverse Events (participants affected / at risk) | 0/53 | 0/70 | 0/59 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Child Pre-visit Prep + Exome (N=53) | Child Pre-visit Prep + Usual Care (N=70) | Child No Pre-visit Prep + Exome (N=59) | Child No Pre-visit Prep + Usual Care (N=68)
Septic Shock (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Disruption of enrollment due to COVID-19 pandemic; required temporary pause in enrollment followed by adjusted study procedures. Instability of study personnel at one enrollment site led to fewer participants enrolled than initially anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (7):
  • Study Protocol (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/Prot_006.pdf
  • Informed Consent Form: 7-14 Assent Form 1 Randomization to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_000.pdf
  • Informed Consent Form: 7-14 Assent Form 2 Assent to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_001.pdf
  • Informed Consent Form: 15-17 Assent Form 1 Randomization to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_002.pdf
  • Informed Consent Form: 15-17 Assent Form 2 Assent to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_003.pdf
  • Informed Consent Form: Consent Form 1 Randomization to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_004.pdf
  • Informed Consent Form: Consent Form 2 Assent to Research (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03548779/ICF_005.pdf